CLINICAL TRIAL: NCT06877572
Title: Enacting Active Survivorship: Implementation of Weight Management Strategies in Endometrial Cancer Survivors
Brief Title: Weight Loss Management in Endometrial Cancer Survivors
Acronym: ECS Weight
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Melissa Javellana, Principal Investigator, University of Kansas Medical Center
Other Study IDs: STUDY00160821
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer Survivors; Weight Management; Early Stage Endometrial Cancer
Keywords: Endometrial Cancer; Endometrial Cancer Survivors; Weight Management; GLP-1 agonist; naltrexone/bupropion; orlistat; phentermine/topiramate
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial cancer survivors with weight management: Survivors of low-risk early-stage endometrial cancer up to 36 months post primary treatment with body mass index (BMI) ≥30 kg/m2
  Interventions: Behavioral: Weight loss with pharmacotherapy; Behavioral: Weight loss without pharmacotherapy

INTERVENTIONS:
Behavioral: Weight loss with pharmacotherapy — Patients will meet with a weight management specialist and discuss their options for weight loss including medications (GLP-1 agonist, naltrexone/bupropion, orlistat, or phentermine/topiramate) or bariatric surgery.
  Other Names: Weight loss medications
Behavioral: Weight loss without pharmacotherapy — Participants not on medications will have their weight recorded at subsequent cancer surveillance or other routine medical visits

SUMMARY:
This study is being done to understand how oncologists can engage a multidisciplinary team to help endometrial cancer survivors with obesity to engage in a weight management program and potentially start a weight loss medication. Obesity often impacts the future health and longevity of early-stage endometrial cancer survivors more than their cancer diagnosis.

Patients will be referred to the KUMC OB/Gyn weight management clinic to discuss weight management options.

* If patients decide to use medications for weight loss, then the study will collect data from their chart that is recorded as part of routine monitoring for patients on weight loss medications.
* If patients decide not to use any medications, the study will monitor physical exam and lab data collected as part of their routine medical care.

The study will also try to understand reasons why patients did or did not start using a weight loss medication.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* ECOG 0-2
* BMI ≥ 30kg/m2
* Completed surgical staging with no evidence of residual disease
* Endometrioid endometrial adenocarcinoma, p53 wild type
* Stage 1
* Undergoing active surveillance +/- brachytherapy

Exclusion Criteria:

* Unable to participate in behavior weight loss
* Stroke, heart attack, end stage liver disease, or end stage kidney disease during the last 6 months.
* Currently on a GLP-1 agonist
* Currently on insulin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors of low-risk early-stage endometrial cancer up to 36 months post primary treatment with body mass index (BMI) ≥30 kg/m^2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants referred to weight loss clinic who are able to start weight management medications | 12 months
  We will track the number of participants who do and do not start medication. Patients will be offered GLP-1 agonist, naltrexone/bupropion, orlistat, or phentermine/topiramate based discussion with weight management specialist.

SECONDARY OUTCOMES:
Change in insulin resistance over 12 months using HgA1c as a surrogate marker in participants on weight loss medications | 12 months
  We will measure HgA1c (%) at baseline and after 6 and 12 months of medication use.
Change in quality of life as assessed by the Functional Assessment of Cancer Therapy- Gynecology (FACT-G) over 12 months in participants on weight loss medications | 12 months
  FACT-G will be assessed at baseline, 6, and 12 months after starting medication. The score ranges from 0-108 with higher scores indicating better quality of life.
Change in depression as assessed by Patient Health Questionnaire-2 (PHQ-2) over 12 months in participants on weight loss medications | 12 months
  PHQ-2 will be assessed at baseline, 6, and 12 months after starting medication. The score ranges from 0-6 with lower scores indicating less depressive symptoms. Patients with a score of 3 or greater will be further assessed with Patient Health Questionnaire-9 and managed per a protocol already in place for all weight loss clinic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial

REFERENCES:
- [Background] Klair N, Patel U, Saxena A, Patel D, Ayesha IE, Monson NR, Ramphall S. What Is Best for Weight Loss? A Comparative Review of the Safety and Efficacy of Bariatric Surgery Versus Glucagon-Like Peptide-1 Analogue. Cureus. 2023 Sep 29;15(9):e46197. doi: 10.7759/cureus.46197. eCollection 2023 Sep. PMID 37905277
- [Background] Tondt, J., et al., Obesity Algorithm eBook, presented by the Obesity Medicine Association. 2023.
- [Background] Eisenberg D, Shikora SA, Aarts E, Aminian A, Angrisani L, Cohen RV, de Luca M, Faria SL, Goodpaster KPS, Haddad A, Himpens JM, Kow L, Kurian M, Loi K, Mahawar K, Nimeri A, O'Kane M, Papasavas PK, Ponce J, Pratt JSA, Rogers AM, Steele KE, Suter M, Kothari SN. 2022 American Society of Metabolic and Bariatric Surgery (ASMBS) and International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) Indications for Metabolic and Bariatric Surgery. Obes Surg. 2023 Jan;33(1):3-14. doi: 10.1007/s11695-022-06332-1. PMID 36336720
- [Background] Lonneman DJ Jr, Rey JA, McKee BD. Phentermine/Topiramate extended-release capsules (qsymia) for weight loss. P T. 2013 Aug;38(8):446-52. PMID 24222976
- [Background] Jain SS, Ramanand SJ, Ramanand JB, Akat PB, Patwardhan MH, Joshi SR. Evaluation of efficacy and safety of orlistat in obese patients. Indian J Endocrinol Metab. 2011 Apr;15(2):99-104. doi: 10.4103/2230-8210.81938. PMID 21731866
- [Background] Kulak-Bejda A, Bejda G, Waszkiewicz N. Safety and efficacy of naltrexone for weight loss in adult patients - a systematic review. Arch Med Sci. 2020 Sep 10;17(4):940-953. doi: 10.5114/aoms.2020.96908. eCollection 2021. PMID 34336024
- [Background] Ussher JR, Drucker DJ. Glucagon-like peptide 1 receptor agonists: cardiovascular benefits and mechanisms of action. Nat Rev Cardiol. 2023 Jul;20(7):463-474. doi: 10.1038/s41569-023-00849-3. Epub 2023 Mar 28. PMID 36977782
- [Background] Gao X, Hua X, Wang X, Xu W, Zhang Y, Shi C, Gu M. Efficacy and safety of semaglutide on weight loss in obese or overweight patients without diabetes: A systematic review and meta-analysis of randomized controlled trials. Front Pharmacol. 2022 Sep 14;13:935823. doi: 10.3389/fphar.2022.935823. eCollection 2022. PMID 36188627
- [Background] Collins L, Costello RA. Glucagon-Like Peptide-1 Receptor Agonists. 2024 Feb 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551568/ PMID 31855395
- [Background] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688
- [Background] Aleksandrova K, Drogan D, Boeing H, Jenab M, Bas Bueno-de-Mesquita H, Jansen E, van Duijnhoven FJ, Rinaldi S, Fedirko V, Romieu I, Kaaks R, Riboli E, Gunter MJ, Romaguera D, Westhpal S, Overvad K, Tjonneland A, Halkjaer J, Boutron-Ruault MC, Clavel-Chapelon F, Lukanova A, Trichopoulou A, Trichopoulos D, Vidalis P, Panico S, Agnoli C, Palli D, Tumino R, Vineis P, Buckland G, Sanchez-Cruz JJ, Dorronsoro M, Diaz MJ, Barricarte A, Ramon Quiros J, Peeters PH, May AM, Hallmans G, Palmqvist R, Crowe FL, Khaw KT, Wareham N, Pischon T. Adiposity, mediating biomarkers and risk of colon cancer in the European prospective investigation into cancer and nutrition study. Int J Cancer. 2014 Feb 1;134(3):612-21. doi: 10.1002/ijc.28368. Epub 2013 Aug 5. PMID 23824948
- [Background] Petersen Harrington S, Balmaceda J, Spoozak L, Jewell A, Fitzgerald-Wolff S. Higher baseline BMI and lower estimated median income associated with increasing BMI after endometrial cancer diagnosis. Gynecol Oncol Rep. 2022 Dec 13;44:101123. doi: 10.1016/j.gore.2022.101123. eCollection 2022 Dec. PMID 36589506
- [Background] Ward KK, Shah NR, Saenz CC, McHale MT, Alvarez EA, Plaxe SC. Cardiovascular disease is the leading cause of death among endometrial cancer patients. Gynecol Oncol. 2012 Aug;126(2):176-9. doi: 10.1016/j.ygyno.2012.04.013. Epub 2012 Apr 13. PMID 22507532
- [Background] Soisson S, Ganz PA, Gaffney D, Rowe K, Snyder J, Wan Y, Deshmukh V, Newman M, Fraser A, Smith K, Herget K, Hanson HA, Wu YP, Stanford J, Al-Sarray A, Werner TL, Setiawan VW, Hashibe M. Long-term Cardiovascular Outcomes Among Endometrial Cancer Survivors in a Large, Population-Based Cohort Study. J Natl Cancer Inst. 2018 Dec 1;110(12):1342-1351. doi: 10.1016/j.ygyno.2017.12.025. PMID 29741696
- [Background] Guh DP, Zhang W, Bansback N, Amarsi Z, Birmingham CL, Anis AH. The incidence of co-morbidities related to obesity and overweight: a systematic review and meta-analysis. BMC Public Health. 2009 Mar 25;9:88. doi: 10.1186/1471-2458-9-88. PMID 19320986
- [Background] Shaw E, Farris M, McNeil J, Friedenreich C. Obesity and Endometrial Cancer. Recent Results Cancer Res. 2016;208:107-136. doi: 10.1007/978-3-319-42542-9_7. PMID 27909905
- [Background] Onstad MA, Schmandt RE, Lu KH. Addressing the Role of Obesity in Endometrial Cancer Risk, Prevention, and Treatment. J Clin Oncol. 2016 Dec 10;34(35):4225-4230. doi: 10.1200/JCO.2016.69.4638. Epub 2016 Nov 7. PMID 27903150
- [Background] Creasman WT. Estrogen and cancer. Gynecol Oncol. 2002 Jul;86(1):1-9. doi: 10.1006/gyno.2001.6499. No abstract available. PMID 12079291
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204